CLINICAL TRIAL: NCT04433351
Title: Evaluation of an Enriched Speech Rehabilitation Program Combining Speech Therapy and Sensory-motor Integration in Aphasic Patients
Brief Title: Sensory-Motor Integration for Speech Rehabilitation in Patients with Post-stroke Aphasia
Acronym: SEMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (Other); GIPSA-LAB (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 38RC20.061; 2020-A00720-39 (Other: ID RCB)
Record Dates: First submitted 2020-05-19; First posted 2020-06-16 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Aphasia Non Fluent; Stroke
Keywords: post-stroke aphasia; non-fluent aphasia; speech rehabilitation; neuroimaging; neural reorganization; recovery
MeSH Terms: conditions — Aphasia, Broca; Stroke

STUDY DESIGN:
Intervention Model Description: Two types of rehabilitation will be compared, a simple rehabilitation (S, based on conventional speech therapy) and an enriched rehabilitation (E, based on the use of sensory-motor integration in addition to conventional speech therapy). The investigators will constitute two cohorts of patients (N=18 per cohort): a cohort SE which will carry out first the simple rehabilitation protocol followed by enriched rehabilitation, and a cohort ES which will carry out first the enriched rehabilitation protocol followed by simple rehabilitation. The protocol starts at T0 (inclusion according to defined criteria) and after a first evaluation (T1), patients will then perform the first part of the rehabilitation protocol during 4 weeks. After these 4 weeks, a second evaluation will be performed (T2). Then, the second part of the rehabilitation protocol will be carried out during 4 weeks. At the end, the T3 evaluation will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SE cohort (Experimental): Patients in the SE cohort will carry out first the simple rehabilitation protocol (S, 4 weeks) followed by enriched rehabilitation (E, 4 weeks).
  Interventions: Device: Enriched rehabilitation; Device: Simple rehabilitation
- ES cohort (Experimental): Patients in the ES cohort will carry out first the enriched rehabilitation protocol (E, 4 weeks) followed by simple rehabilitation (S, 4 weeks).
  Interventions: Device: Enriched rehabilitation; Device: Simple rehabilitation

INTERVENTIONS:
Device: Enriched rehabilitation — The enriched rehabilitation is based on the use of sensory-motor integration in addition to conventional speech therapy. The sensory-motor integration method is based on the Ultraspeech-player software. This software allows therapists to display movements of speech articulators (tongue and lips) recorded on a reference speaker during production of vowels or consonants (isolated or combined). Sagittal movements of the tongue are recorded using ultrasound and front views of lip movements are captured through video imaging.
  During rehabilitation with the Ultraspeech-player software, patients will be seated in front of a computer screen, observe articulatory movements and listen to phonemes. Then, they will be required to repeat each of them five times and move on to the next phoneme, with the agreement of the experimenter.
  Other Names: Sensory-motor integration; Illustration-based rehabilitation method
Device: Simple rehabilitation — The simple rehabilitation is based on conventional speech therapy. The conventional speech therapy will be provided by the speech therapist. Classically, the speech therapist uses word production with repetition and naming exercises. The therapist will show the patient series of pictures associated or not with written words, and the patient is required to name them and/or read aloud the word. In case of impossibility to perform the task, the therapist may can help the patient by using the indexing method or by asking the patient to repeat after him/her. According to patient's competencies and progress, the difficulty of reeducation can increase progressively.
  Other Names: Conventional speech therapy

SUMMARY:
SEMO is a multidisciplinary project (language sciences, cognitive psychology and neuropsychology, physical medicine and rehabilitation, neurology, speech-language pathology, functional neuroimaging and engineering sciences) that aims first, to test and develop a novel speech rehabilitation program designed for patients with non-fluent aphasia and, second, to better describe neural reorganization after successful recovery. To this end, the investigators will conduct a prospective monocentric cross-over study, including two cohorts of post-stroke aphasic patients and two control groups.

DETAILED DESCRIPTION:
In this project, the investigators propose to evaluate the effectiveness of a new rehabilitation program, based on illustration of speech articulators, to improve speech in patients with non-fluent aphasia. The instigators' method is based on the reinforcement of the interaction between perceptual and motor representations, thanks to the innovative Ultraspeech device. The investigators will exploit a fundamental psycholinguistic principle, which postulates that speech is based both on the activation of the system controlling the motricity of effectors related to word articulation (action) and on the auditory or visual representation of words (perception). The sensory-motor interaction method that the investigators propose allows the patient to perceive phonemes and visualize on a computer screen the movements of the tongue and lips previously recorded by a healthy speaker, typically a speech therapist. Through repeated exercises, the patient is trained to produce sounds correctly, using the correct pronunciation and articulatory movements of the reference speaker as a model. The investigators will compare patients who will follow a classical speech and language therapy rehabilitation program followed by an 'enriched' rehabilitation program including rehabilitation based on sensory-motor interaction associated with speech and language therapy, and vice versa. In order to judge the favorable effect of the rehabilitation program including sensory-motor integration, the following measures will be considered: (a) language skills, (b) phonemic quality, (c) inner speech abilities and (d) cognitive function. Brain language networks will be evaluated with neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-fluent aphasia after lesion in the dominant hemisphere for language
* native speakers of French
* normal or corrected to normal vision
* satisfying all criteria for the MRI examination

Exclusion Criteria:

* patients with comprehension deficits, hemi-spatial neglect or upper limb apraxia

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of acoustic changes in the speech signal before and after each rehabilitation protocol | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of acoustic properties (formants, voice onset time and spectral moments) with a phoneme repetition task. Repeated phonemes are isolated vowels, semi-consonants in vowel context and consonants in /a/ context with the consonants (C) placed in initial (/Ca/) or medial (/aCa/) positions.

SECONDARY OUTCOMES:
Evaluation of changes in inner speech abilities before and after each rehabilitation protocol - Inner speech testing 1 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Evaluate inner speech abilities with an introspective questionnaire
Evaluation of changes in inner speech abilities before and after each rehabilitation protocol - Inner speech testing 2 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Evaluate inner speech abilities with a behavioral task (homophone detection task)
Clinical language assessment 1a | Baseline pre-intervention
  Assessment of oral and written expression with BDAE (Boston Diagnostic Aphasia Examination).
Evaluation of changes in language abilities before and after rehabilitation - Clinical language assessment 1b | Immediately after the first intervention; immediately after the second intervention
  Assessment of oral expression (picture naming) with BDAE (Boston Diagnostic Aphasia Examination).
Clinical language assessment 2a | Baseline pre-intervention
  Assessment of transcoding (word/sentence repetition and syllable/word reading) with BDAE (Boston Diagnostic Aphasia Examination).
Evaluation of changes in language abilities before and after rehabilitation - Clinical language assessment 2b | Immediately after the first intervention; immediately after the second intervention
  Assessment of transcoding (word repetition and word reading) with BDAE (Boston Diagnostic Aphasia Examination).
Evaluation of changes in language abilities before and after each rehabilitation protocol - Clinical language assessment 3 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of verbal fluency with phonemic and semantic fluency tasks. The patient must generate words that satisfy certain criteria: beginning with a particular letter (phonemic fluency) or belonging to a particular semantic category (semantic fluency).
Clinical language assessment 4 | Baseline pre-intervention
  Assessment of bucco-facial praxia with MT-86 (Montreal-Toulouse aphasia language examination protocol).
Evaluation of changes in language abilities before and after each rehabilitation protocol - Clinical language assessment 5 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of phonemic discrimination with BALE (Batterie Analytique du Langage Ecrit).
Evaluation of changes in language abilities before and after each rehabilitation protocol - Clinical language assessment 6 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of phonological awareness with a rhyme detection task. The patient must decide whether two heard words rhyme or not.
Evaluation of changes in cognitive level before and after each rehabilitation protocol - Neuropsychological assessment 1 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of general cognitive level with CASP (Cognitive Assessment Scale for Stroke Patients). CASP evaluates several abilities (naming, comprehension, inhibition, flexibility etc.) and the global score is out of 36.
Evaluation of changes in specific executive functions before and after each rehabilitation protocol - Neuropsychological assessment 2 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of visuo-spatial span with the Corsi blocks task.
Evaluation of changes in specific executive functions before and after each rehabilitation protocol - Neuropsychological assessment 3 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of non-verbal fluency with the Ruff figural fluency test.
Evaluation of changes in specific executive functions before and after each rehabilitation protocol - Neuropsychological assessment 4 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of executive functions with the TMT A-B (Trail Making Test A-B).
Evaluation of changes in non-verbal episodic memory before and after each rehabilitation protocol - Neuropsychological assessment 5 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of non-verbal episodic memory with BEM84 (Batterie d'Efficience Mnésique de Signoret). This test contains an immediate recall task (score out of 12) and a delayed recall task (score out of 12).
Evaluation of changes in mental rotation abilities before and after each rehabilitation protocol - Neuropsychological assessment 6 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of mental rotation abilities.
Evaluation of mood changes before and after each rehabilitation protocol - Neuropsychological assessment 7 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of depression with Aphasic Depression Rating Scale (ADRS; score out of 32; a score lower than 7 is for "no depression").
Evaluation of mood changes before and after each rehabilitation protocol - Neuropsychological assessment 8 | Baseline pre-intervention; immediately after the first intervention; immediately after the second intervention
  Assessment of anxiety with Hamilton scale (score out of 56; a score lower or equal to 12 is for "normal anxiety"; a score between 12 and 20 is for "mild anxiety"; a score between 20 and 25 is for "moderate anxiety"; a score higher than 25 is for "severe anxiety").
Neuropsychological assessment 9 | Baseline pre-intervention
  Assessment of familiarity degree with digital tools with an in-house test developed by the neuropsychologists from our clinical setting. This task allows to evaluate the use of the computer tools, its frequency of use and the type of activities carried out.
Evaluation of brain network activation (with measurement of BOLD, Blood Oxygen Level Dependent) before and after rehabilitation - Evaluation-brain 1 | Baseline pre-intervention; immediately after the first intervention
  Assessment of brain networks modulation with fMRI (functional MRI) tasks : syllable repetition (repeating a heard syllable), picture-prompted rhyme detection (judging if verbal labels of pictures presented in pairs rhyme or not), and picture naming (naming pictures).
Evaluation of brain functional connectivity before and after rehabilitation - Evaluation-brain 2 | Baseline pre-intervention; immediately after the first intervention
  Assessment of functional connectivity with rs-fMRI (resting state-functional MRI).
Evaluation of brain anatomical connectivity before and after rehabilitation - Evaluation-brain 3 | Baseline pre-intervention; immediately after the first intervention
  Assessment of diffuse white-matter changes in multiple bundles with MRI-DTI (Diffusion Tension Imaging).

CONTACTS AND LOCATIONS:
Overall Officials: Monica Baciu, MD PhD, Principal Investigator — University Hospital, Grenoble & Laboratoire de Psychologie et NeuroCognition
Locations (1):
- Chu Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No